CLINICAL TRIAL: NCT00480454
Title: An Open Randomized Dose Selection Study Evaluating the Safety, Immunogenicity, and Impact of a TB Vaccine, MVA85A, on the Immunogenicity of EPI Vaccines Administered Simultaneously to Healthy Infants Previously Vaccinated With BCG.
Brief Title: Safety, Immunogenicity, and Impact of MVA85A, on the Immunogenicity of the EPI Vaccines
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Dr Helen McShane, University of Oxford
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TB012
Record Dates: First submitted 2007-05-30; First posted 2007-05-31 (Estimated); Last update posted 2010-02-09 (Estimated); Status verified 2010-02

CONDITIONS: TB
Keywords: TB; Tuberculosis; Infants; EPI
MeSH Terms: conditions — Tuberculosis | interventions — MVA 85A; MVA Pfs25-IMX313 malaria vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Stage 1 would require 12 per group low dose and 12 per group high dose (total 72)
  Interventions: Biological: MVA 85A
- 2 (Active Comparator): Stage 2 would require 48 per group (total 144)
  Interventions: Biological: MVA 85A

INTERVENTIONS:
Biological: MVA 85A — intradermal vaccine
  Other Names: TB vaccine; modified vaccinia virus Ankara

SUMMARY:
This study is preliminary to proving that this vaccine could protect against tuberculosis in humans. Although there is no proven data to show that infants will benefit directly from participation in this study by being protected against TB, MVA85A protection of mice, guinea pigs and monkeys against tuberculosis is encouraging. It is hoped that the information gained from this study will contribute to the development of a safe and effective TB vaccine for HIV negative and positive individuals. Participants in this study will benefit by having information about their general health status, and the rigorous follow up visit that could enhance early detection and management of medical conditions that might arise in the course of the study.

DETAILED DESCRIPTION:
Over the last 3 years Phase I studies with MVA85A allowed for sequential vaccination of volunteer groups with a step-wise increase in mycobacterial exposure, to minimize the possibility of a Koch reaction. Trials were also conducted sequentially in the UK and The Gambia, as there is a greater degree of exposure to both environmental mycobacteria and M.tb in The Gambia. A Koch reaction describes the development of immunopathology in a person or animal with tuberculosis, when an exaggerated immune response to M.tb is stimulated. It has now been demonstrated in the mouse model of therapeutic vaccination (Taylor et al, 2003). Available animal data suggest that these reactions do not occur in mice latently infected with M.tb, suggesting that such reactions may correlate with high bacterial load and that the Koch phenomenon may not pose a problem for vaccination of healthy albeit latently infected humans (Taylor et al, 2003).

In the UK, 14 mycobacterially and BCG naïve, healthy volunteers were vaccinated twice with 5 x 107pfu MVA85A, administered intradermally at 3 week intervals. MVA85A was found to be safe and well tolerated. A single vaccination with MVA85A induced remarkably high levels of specific effector T cell responses 1 week after vaccination (mean γ IFN Elispot response to PPD was 460 spots per million PBMC). MVA85A was also safe in 17 volunteers vaccinated with BCG in the previous 0.5-37 years. The safety profile of MVA85A in these 17 volunteers was the same as in the BCG naïve group. Interestingly, these 17 volunteers showed even higher peak levels of antigen specific T cells (mean response to PPD was 917 spots per million PBMC) 1 week post-vaccination than those immunized with MVA85A alone. Perhaps more importantly for the induction of T cell memory, these volunteers who were previously BCG vaccinated maintained significantly higher levels of antigen specific T cells after MVA85A for up to 24 weeks after vaccination, when compared to those volunteers vaccinated with either BCG or MVA85A alone (McShane et al, 2004). The next trial in the UK looked at the boosting efficacy of MVA85A when administered one month after BCG vaccination. 10 healthy, BCG naïve volunteers were vaccinated with BCG and one month later were boosted with MVA85A. Safety and boosting efficacy was comparable to the previous trial where the interval between BCG and MVA85A was 0.5-37 years.

2.3.2 Gambian studies Following the success of the trials with MVA85A in the UK, a collaboration with the MRC unit in The Gambia was initiated. MVA85A was first evaluated in Phase I clinical trials in BCG naïve subjects (n = 11) and subsequently in BCG primed subjects (n=10). In these studies the safety and immunogenicity profile is comparable to that seen in the UK studies. In both the UK and The Gambian studies, MVA85A induces 5-10 fold higher immune responses than any other recombinant MVA in clinical trials. The most likely explanation for this is that the volunteers have some weak pre-existing anti-mycobacterial immunity induced by exposure to environmental mycobacteria, and this is being boosted by vaccination with MVA85A. When MVA85A is administered to BCG naïve subjects in the Gambia, the magnitude and kinetics of response resemble the BCG primed group in the UK, a finding that is likely to represent a greater degree of environmental priming in tropical climates.

Taken together, over 600 people, including HIV positive and over 250 Gambian adults and children, have now been immunised with various recombinant MVA investigational vaccines including constructs expressing malaria, HIV, hepatitis B and melanoma antigens without significant adverse reactions (Hill, unpublished data). Furthermore, 190 children aged 1-5 years were vaccinated with a recombinant MVA expressing a malarial antigen in 2006, with no vaccine related SAEs (Hill, personal communication). This safety data now allows for progression to testing MVA85A in a phase II study in infants who have been vaccinated with BCG, in a Gambian population which may include low numbers of latently M.tb infected and HIV positive children.

It is important to test the safety, immunogenicity, and possible interference (detrimental, none or beneficial) with other EPI vaccines of the MVA85A vaccine in such a group, which is one of the potential target populations for a large-scale efficacy study. Also the effects of simultaneous EPI vaccine administration on the immunogenicity of MVA85A need to be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants aged 2 - 3 months
* Recorded BCG vaccination within first two weeks of life with typical BCG scar on the left arm
* Receiving standard EPI immunizations according to national immunization programme (DTwPHib at 2/3/4 months, OPV at birth, 1, 2 and 3 months, Hep B at birth, 2 & 4 months)
* Written informed consent by parent / guardian

Exclusion Criteria:

* Any clinically significant abnormal finding on screening from biochemistry or haematology
* Any AIDS defining illness
* Prior receipt of a recombinant MVA or Fowlpox vaccine, or other experimental vaccine
* Use of any investigational or non-registered drug, live vaccine or medical device other than the study vaccine within 2 weeks preceding dosing of study vaccine, or planned use during the study period
* Administration of chronic (defined as more than 14 days) immunosuppressive drugs or other immune modifying drugs within 6 months of vaccination. (For corticosteroids, this will mean prednisolone, or equivalent, ≥ 0.5 mg/kg/day. Inhaled and topical steroids are allowed.)
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, e.g. egg products
* Presence of any underlying disease that compromises the diagnosis and evaluation of response to the vaccine
* History of > 2 hospitalisations for invasive bacterial infections (pneumonia, meningitis)
* Any other on-going chronic illness requiring hospital specialist supervision
* Administration of immunoglobulins and/or any blood products within one month preceding the planned administration of the vaccine candidate
* Any history of anaphylaxis in reaction to vaccination
* Research Physician's assessment of lack of willingness by parents to participate and comply with all requirements of the protocol, or identification of any factor felt to significantly increase the infant's risk of suffering an adverse outcome
* Likelihood of travel away from the study area
* Untreated malaria infection

Ages: 2 Months to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 214 (Actual)
Dates: Start 2006-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Dose selection, safety and immunogenicity of MVA85A vaccines in 4 month old healthy Gambian infants | one year

SECONDARY OUTCOMES:
Impact of MVA85A on the immunogenicity of EPI vaccines (DTwPHib, Hep B) and vice versa when administered simultaneously to children who have had BCG vaccine within the first two weeks of life. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Helen McShane, Principal Investigator — University of Oxford
Locations (1):
- MRC, Banjul, The Gambia

REFERENCES:
- [Background] McShane H, Pathan AA, Sander CR, Keating SM, Gilbert SC, Huygen K, Fletcher HA, Hill AV. Recombinant modified vaccinia virus Ankara expressing antigen 85A boosts BCG-primed and naturally acquired antimycobacterial immunity in humans. Nat Med. 2004 Nov;10(11):1240-4. doi: 10.1038/nm1128. Epub 2004 Oct 24. PMID 15502839
- [Background] Goonetilleke NP, McShane H, Hannan CM, Anderson RJ, Brookes RH, Hill AV. Enhanced immunogenicity and protective efficacy against Mycobacterium tuberculosis of bacille Calmette-Guerin vaccine using mucosal administration and boosting with a recombinant modified vaccinia virus Ankara. J Immunol. 2003 Aug 1;171(3):1602-9. doi: 10.4049/jimmunol.171.3.1602. PMID 12874255
- [Background] Bejon P, Peshu N, Gilbert SC, Lowe BS, Molyneux CS, Forsdyke J, Lang T, Hill AV, Marsh K. Safety profile of the viral vectors of attenuated fowlpox strain FP9 and modified vaccinia virus Ankara recombinant for either of 2 preerythrocytic malaria antigens, ME-TRAP or the circumsporozoite protein, in children and adults in Kenya. Clin Infect Dis. 2006 Apr 15;42(8):1102-10. doi: 10.1086/501459. Epub 2006 Mar 14. PMID 16575727
- [Background] Huygen K, Content J, Denis O, Montgomery DL, Yawman AM, Deck RR, DeWitt CM, Orme IM, Baldwin S, D'Souza C, Drowart A, Lozes E, Vandenbussche P, Van Vooren JP, Liu MA, Ulmer JB. Immunogenicity and protective efficacy of a tuberculosis DNA vaccine. Nat Med. 1996 Aug;2(8):893-8. doi: 10.1038/nm0896-893. PMID 8705859